CLINICAL TRIAL: NCT02757378
Title: A Randomized Controlled Trial of Manual Therapy as a Form of Sensory Discrimination in Chronic Low Back Pain
Brief Title: Manual Therapy as a Form of Sensory Discrimination in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Farrell (Other)
Responsible Party: Sponsor-Investigator, Kevin Farrell, Professor and Chair, Clinical Residency Program in Orthopaedic Physical Therapy, St. Ambrose University
Organization: St. Ambrose University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StAmbroseU
Record Dates: First submitted 2016-04-12; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Low Back Pain
Keywords: Pain; Brain; Plasticity; Education; Manual Therapy; Straight Leg Raise; Remapping
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuroplasticity Education Group (Experimental): Patients who receive manual physical therapy treatment with a neuroplasticity explanation of the basis for the technique
  Interventions: Procedure: Neuroplasticity Explanation (Experimental)
- Biomechanical Education Group (Active Comparator): Patients who receive manual physical therapy treatment with a traditional, biomechanical explanation of the basis for the technique
  Interventions: Procedure: Biomechanical Explanation (Control)

INTERVENTIONS:
Procedure: Neuroplasticity Explanation (Experimental) — Patients were given an explanation of how the brain uses the information from a manual therapy technique to help it remain sharp in identifying where this input is coming from.
  Arms: Neuroplasticity Education Group
Procedure: Biomechanical Explanation (Control) — Patients were given an explanation of how the manual therapy technique affects the anatomy and physiology of the back.
  Arms: Biomechanical Education Group

SUMMARY:
This study evaluates whether different explanations given to patients with long lasting back pain influence a physical therapy treatment technique. Half of the patients will receive an explanation of the proposed treatment technique focusing on how their joints are moving and not moving. The second half of the group will receive the same treatment technique as the first group, but their explanation of the technique's purpose will focus on how their brain interprets the information. The study aims to determine if patients have a different response to the treatment based on the words chosen to explain the technique.

DETAILED DESCRIPTION:
Traditional treatment provided by physical therapists to patients with chronic low back pain focuses on the biomechanical or anatomical impact to local tissues. Recent research has shown that treatment effects may be more related to the understanding of the structural and functional changes in the brain of someone suffering from chronic low back pain. This research implicates that the patients understanding and interpretation of input to the brain may change the patient's perceived representation and interpretation of output of pain within the brain.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18
* Presenting at Physical Therapy with a primary complaint of Low Back Pain
* Low Back Pain being present for 6 months or more
* Fluent in English and willing to participate in the study.

Exclusion Criteria:

* Medical precautions to the use of manual therapy (metal, skin lesions, etc.)
* Prior spine surgery
* Unable to lay prone for the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Low back pain rating change | Within a single, one hour session
  Change, measured within a single, one hour session, of baseline measurements taken, followed immediately by the education / treatment, followed immediately by post-education / treatment measurement of the patient's pain in low back on a numeric pain rating scale of 0 to 10
Leg pain rating | Within a single, one hour session
  Change, measured within a single, one hour session, of baseline measurements taken, followed immediately by the education / treatment, followed immediately by post-education / treatment measurement, level of patient's leg pain on a numeric pain rating scale of 0 to 10.
Active trunk forward flexion | Within a single, one hour session
  Change, measured within a single, one hour session, of baseline measurements taken, followed immediately by the education / treatment, followed immediately by post-education / treatment measurement of distance from longest finger to the floor when patient bends forward (in cm).
Straight Leg Raise | Within a single, one hour session
  Change, measured within a single, one hour session, of baseline measurements taken, followed immediately by the education / treatment, followed immediately by post-education / treatment measurement of angle to which the patient's most affected leg can be lifted (measured in degrees using an inclinometer).

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Louw, PT, PhD, Principal Investigator — International Spine Pain Institute
Locations (5):
- United States (5):
  - Rock Valley Physical Therapy, Moline, Illinois
  - Rock Valley Physical Therapy, Silvis, Illinois
  - Edward Health & Fitness Center & Spa at Seven Bridges, Woodridge, Illinois
  - Rock Valley Physical Therapy, Davenport, Iowa
  - Genesis Physical Therapy and Sports Medicine, Davenport, Iowa

IPD SHARING:
Plan to Share IPD: No